CLINICAL TRIAL: NCT02864446
Title: The Clinical Utility of Urine Intestinal Fatty Acid Binding Protein in the Management of Very Low Birth Weight Infants With Meconium Obstruction
Brief Title: Intestinal Fatty Acid Binding Protein in Very Low Birth Weight Infants With Meconium Obstruction
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Professor, Seoul National University Hospital
Other Study IDs: 1208-071-422
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Meconium Obstruction of Prematurity
MeSH Terms: conditions — Meconium Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Urinary intestinal fatty acid binding protein (i-FABP), a marker of intestinal mucosal cell damage, has recently been proposed as a clinically useful measure in the early detection of necrotizing enterocolitis (NEC). However, there are no data on urinary i-FABP in meconium obstruction of prematurity (MOP). This study aimed to evaluate urinary i-FABP in MOP patient as a marker for early detection.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants weighing <1,250g

Exclusion Criteria:

* major congenital anomalies
* perinatal asphyxia (cord pH <7.0)

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants weighing <1,250g who were admitted in neonatal intensive care unit at Seoul National University Children's Hospital
  * Initial urine samples are collected at the time of 12, 24, 48 hours (+/- 6 hours) after birth.
  * Further urine samples are collected every 48 hours when the enteral feeding starts. (till the amount of feeding reaches to 40mL/kg/day)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comparison of i-FABP level between the meconium obstruction group and the normal feeding advance group | within 48 hours after birth

OTHER OUTCOMES:
Comparison of i-FABP level between breast milk feeding and formular feeding in the normal feeding advance group | through study completion (an average of 1 month)
Comparison of i-FABP level between preterm infants with small for gestational age and without small for gestational age in the normal feeding advance group | within 48 hours after birth
Comparision of i-FABP level between preterm infants with chorioamnionitis and without chorioamnionitis in the normal feeding advance group | within 48 hours after birth
Comparision of i-FABP level between preterm infants with maternal pregnancy induced hypertension (PIH) and without maternal PIH in the normal feeding advance group | within 48 hours after birth
Comparison of i-FABP level between preterm infants with maternal premature rupture of membrane (PROM) and without PROM in the normal feeding advance group | within 48 hours after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes